CLINICAL TRIAL: NCT05776030
Title: Multi-speed Ergonomic Wheelchair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3664-R; 1 I02 RX003664-01P2 (Other Grant/Funding Number: RR&D)
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Diseases; Spinal Cord Injuries
Keywords: Wheelchairs; Community Participation; Social Participation; Ergonomics; Self-Help Devices
MeSH Terms: conditions — Spinal Cord Diseases; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: H1) Single group assignment with crossover design where participant will be randomized which of 3 gear ratios they start with and then which is second, than the last one. n=18
  H2) Two Groups for randomized assignment of which chair (geared or not) the participant starts with and then crosses over to second chair. n=12
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Ergonomic Wheelchair Gear Testing (Experimental): This study has two aims. The first aim will have participants use a single speed ergonomic wheelchair to test three different gear ratio set ups (3:2, 1:1, 2:3).
  Interventions: Device: Single Speed Ergonomic Wheelchair
- Multispeed Testing - Ergonomic Wheelchair (Experimental): The second aim will have participants compared to the participant's standard wheelchair to a multi-speed (2 gear ratios) ergonomic wheelchair.
  Interventions: Device: Multi-Speed Ergonomic Wheelchair
- Multispeed Testing - Standard Wheelchair (Experimental): The second aim will have participants compared to the participant's standard wheelchair to a multi-speed (2 gear ratios) ergonomic wheelchair.
  Interventions: Device: Multi-Speed Ergonomic Wheelchair

INTERVENTIONS:
Device: Single Speed Ergonomic Wheelchair — Ergonomic wheelchair. The ergonomic wheelchair was developed by the MADE program and has anterior placed hand rims that are connected with a bicycle chain. In Aim 1, Participants will use the ergonomic wheelchair to test 3 different gear ratios.
  1. 2:3
  2. 1:1
  3. 3:2
  Arms: Ergonomic Wheelchair Gear Testing
Device: Multi-Speed Ergonomic Wheelchair — The multi-speed ergonomic wheelchair will be developed by the MADE program and will use a two-hand rim design so the participant can change gears by changing hand rims.
  Arms: Multispeed Testing - Ergonomic Wheelchair; Multispeed Testing - Standard Wheelchair

SUMMARY:
Over one million Americans rely on their upper extremities for manual wheelchair propulsion. Shoulder overuse injuries are prevalent among manual wheelchair users and these injuries often result in shoulder pain. Severe shoulder pain can lead some wheelchair users to transition from manual to powered mobility, complicating transportation, and reducing independence in activities of daily living. This project will expand the understanding of a new wheelchair design that allows better positioning of the hand rims and allows for different gearing. The investigators will study steady-state propulsion efficiency with different gear ratios and develop a new system with multiple gear ratios. The advanced gearing will allow for a low gear when initiating movement, going uphill, or when moving over carpet, and then a higher gear option for movements on hard flat level terrain. This system has the potential to dramatically improve shoulder ergonomics and reduce pain in many future manual wheelchair users.

DETAILED DESCRIPTION:
The Minneapolis Adaptive Design & Engineering (MADE) Program has recently developed ergonomic wheelchairs that use a chain drive system to place the hand rims in an ergonomic position while keeping the rear drive wheels posterior for a stable base of support. The investigators' ergonomic wheelchair's forward hand rim positioning allows for a more efficient push along a longer arc length of the hand rims, without sacrificing wheelchair stability or shoulder ergonomics.

The ergonomic wheelchair's chain drive allows for individualized gear ratios to suit each wheelchair user's needs; however, the investigators have not yet studied this feature. Thus, the objectives of this proposed work are to (1) explore the effect of different gearing options on Veteran wheelchair user steady-state propulsion efficiency, and (2) develop a multi-speed ergonomic wheelchair allowing for lower gears during difficult situations (initiating movements, moving over carpeting) and higher gears for steady-state movements on flat surfaces.

The investigators will recruit 18 Veterans with SCI/D to participate in a cross-over study of the ergonomic wheelchair with three gear ratios (3:2 (low), 1:1 (normal), and 2:3 (high)). The investigators will use two measurement approaches to assess efficiency: (1) work done at the pushrim hubs to move the wheelchair in Joules (J), and (2) the measurement of energy (kCal: kilocalories) expended by the Veteran to move the wheelchair. Similar to miles per gallon in a car, the investigators will calculate distances traveled in meters (m) per energy units (m/J and m/kCal) as the measures of efficiency. The investigators hypothesize that (H1) Higher gear ratios will be more efficient (higher m/J) on hard level terrain than lower gear ratios, (H2) Lower gear ratios will be more efficient (higher m/J) for inclined terrain than higher gear ratios, (H3) Lower gear ratios will be more efficient (higher m/J) for carpeted terrain than higher gear ratios, and (H4) Veterans will be more efficient (higher m/kCal) in moving the wheelchair during the 6MPT on hard level terrain when using higher gear ratios compared with lower gear ratios. In addition to steady-state measures, the investigators will also explore the effects of gearing on propulsion initiation and expect lower gear ratios will be beneficial for initiation on all terrains.

The investigators will then recruit 12 Veterans to try a new multi-speed ergonomic wheelchair that has two hand rims per side - one in a lower gear and the other in a higher gear. The proposed system does not require manual or electric shifting between gears. Instead, the Veteran can use the lower gear to initiate movements and then "shift on the fly" by simply pushing on the other hand rim. Veterans will return to the laboratory and provide feedback as the design is iteratively improved. Quantitative and qualitative data will be captured to determine feasibility of this approach and to promote commercialization of the multi-speed ergonomic wheelchair.

Throughout the project, the team will work closely with VA's Technology Transfer Program and the TechLink Center to find an industry partner for this work. The investigators' team has demonstrated the ability to develop rehabilitation products into commercially licensed products. The investigators will follow a similar stage-gate process in this development project to maximize the chances for successful commercialization of the modular multi-speed ergonomic wheelchair.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Uses manual wheelchair daily
* Mass less than 125 kg
* Age 18 or older
* Decisional competency to provide consent and cognitive ability to participate fully in study procedures
* Body size appropriate to fit the wheelchairs (16" and 18" seat widths)

Exclusion Criteria:

Exclusion criteria:

* Sitting surface pressure injuries
* Flap procedure to address pressure injury less than one year earlier
* Unable to obtain clinically acceptable seating system for study wheelchairs
* Not able to propel a manual wheelchair
* Upper extremity or spine issues which would make this study unsafe, such as recent surgeries, fractures, tendon tears or nerve impingement (will be assessed by SCI physician - Dr. Byron Eddy)
* Medical conditions such as cardiovascular disease, pulmonary disease, or other conditions that would make the study procedures unsafe (will be assessed by SCI physician - Dr. Byron Eddy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
20 Meter Push Test - level surface, Gear Ratio 1:1 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - level surface, Gear Ratio 2:3 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - level surface, Gear Ratio 3:2 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - uphill, Gear Ratio 1:1 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - uphill, Gear Ratio 2:3 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - uphill, Gear Ratio 3:2 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - Carpet, Gear Ratio 1:1 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - Carpet, Gear Ratio 2:3 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
20 Meter Push Test - Carpet, Gear Ratio 3:2 | up to 4 weeks after enrollment
  Individuals self-propel a wheelchair 20 meters at their chosen pace
6 Minute Push Test - Usual Wheelchair, Temporal/Spatial | up to 4 weeks after enrollment
  Distance (m) and number of pushes will be collected during this test.
6 Minute Push Test - Gear Ratio 1:1, Temporal/Spatial | up to 4 weeks after enrollment
  Distance (m) and number of pushes will be collected during this test.
6 Minute Push Test - Gear Ratio 2:3, Temporal/Spatial | up to 4 weeks after enrollment
  Distance (m) and number of pushes will be collected during this test.
6 Minute Push Test - Gear Ratio 3:2, Temporal/Spatial | up to 4 weeks after enrollment
  Distance (m) and number of pushes will be collected during this test.
6 Minute Push Test - Usual Wheelchair, Metabolic (kCal/min) | up to 4 weeks after enrollment
  Oxygen Uptake (VO2: L/min), Carbon dioxide production (VCO2: L/min), and respiratory quotient (RQ) will all be collected using a COSMED K5 portable metabolic measurement system
  These measures are used for calculating kCal/min = ([1.1 * RQ] + 3.9) * VO2
6 Minute Push Test - Gear Ratio 1:1, Metabolic (kCal/min) | up to 4 weeks after enrollment
  Oxygen Uptake (VO2: L/min), Carbon dioxide production (VCO2: L/min), and respiratory quotient (RQ) will all be collected using a COSMED K5 portable metabolic measurement system
  These measures are used for calculating kCal/min = ([1.1 * RQ] + 3.9) * VO2
6 Minute Push Test - Gear Ratio 2:3, Metabolic (kCal/min) | up to 4 weeks after enrollment
  Oxygen Uptake (VO2: L/min), Carbon dioxide production (VCO2: L/min), and respiratory quotient (RQ) will all be collected using a COSMED K5 portable metabolic measurement system
  These measures are used for calculating kCal/min = ([1.1 * RQ] + 3.9) * VO2
6 Minute Push Test - Gear Ratio 3:2, Metabolic (kCal/min) | up to 4 weeks after enrollment
  Oxygen Uptake (VO2: L/min), Carbon dioxide production (VCO2: L/min), and respiratory quotient (RQ) will all be collected using a COSMED K5 portable metabolic measurement system
  These measures are used for calculating kCal/min = ([1.1 * RQ] + 3.9) * VO2
Wheelchair Skills Test Version 5.2 - Usual Wheelchair | up to 4 weeks after enrollment
  The WST is used for objective evaluation of manual wheelchair skills. It includes 32 skills that are rates advanced pass/highly proficient (3 points), pass (2 points), pass with difficulty (1 point), or fail (0 points). The WST covers a wide variety of skills that manual wheelchair users experience in everyday life including inclines, side slopes, soft surface, thresholds, gaps, curbs, obstacle avoidance, and wheelies.
Wheelchair Skills Test Version 5.2 - Multispeed Wheelchair | up to 4 weeks after enrollment
  The WST is used for objective evaluation of manual wheelchair skills. It includes 32 skills that are rates advanced pass/highly proficient (3 points), pass (2 points), pass with difficulty (1 point), or fail (0 points). The WST covers a wide variety of skills that manual wheelchair users experience in everyday life including inclines, side slopes, soft surface, thresholds, gaps, curbs, obstacle avoidance, and wheelies.
600 Meter Course - Usual Wheelchair, Timed (seconds) | up to 4 weeks after enrollment
  The distance of 600 meters is used clinically to assess community ambulation ability and can be used to determine if a power wheelchair is needed. The 600 meter course will include several turns, carpeting, and starting/stopping the wheelchair.
  Participants will be instructed to complete the course at a comfortable pace and will be timed (s).
600 Meter Course - Multispeed Wheelchair, Timed (seconds) | up to 4 weeks after enrollment
  The distance of 600 meters is used clinically to assess community ambulation ability and can be used to determine if a power wheelchair is needed. The 600 meter course will include several turns, carpeting, and starting/stopping the wheelchair.
  Participants will be instructed to complete the course at a comfortable pace and will be timed (s).
600 Meter Course - Usual Wheelchair, Rating of Perceived Exertion (RPE) | up to 4 weeks after enrollment
  The distance of 600 meters is used clinically to assess community ambulation ability and can be used to determine if a power wheelchair is needed. The 600 meter course will include several turns, carpeting, and starting/stopping the wheelchair.
  Participants will be instructed to complete the course at a comfortable pace and RPE will be asked at the end of the course.
600 Meter Course - Multispeed Wheelchair, Rating of Perceived Exertion (RPE) | up to 4 weeks after enrollment
  The distance of 600 meters is used clinically to assess community ambulation ability and can be used to determine if a power wheelchair is needed. The 600 meter course will include several turns, carpeting, and starting/stopping the wheelchair.
  Participants will be instructed to complete the course at a comfortable pace and RPE will be asked at the end of the course.
Mobility-Related ADL - Usual Wheelchair, Timed (seconds) | up to 4 weeks after enrollment
  This is a standardized, timed circuit of simulated mobility-related ADL tasks to simulate a morning ADL routine.
Mobility-Related ADL - Multispeed Wheelchair, Timed (seconds) | up to 4 weeks after enrollment
  This is a standardized, timed circuit of simulated mobility-related ADL tasks to simulate a morning ADL routine.
Mobility-Related ADL - Usual Wheelchair, Independency | up to 4 weeks after enrollment
  This is a standardized, timed circuit of simulated mobility-related ADL tasks to simulate a morning ADL routine. All ICF activity-based measures of function in a wheelchair. Independence for tasks will be scored using the Function Everyday with a Wheelchair Capacity scoring from 0 (dependent) to 3 (independent).
Mobility-Related ADL - Multispeed Wheelchair, Independency | up to 4 weeks after enrollment
  This is a standardized, timed circuit of simulated mobility-related ADL tasks to simulate a morning ADL routine. All ICF activity-based measures of function in a wheelchair. Independence for tasks will be scored using the Function Everyday with a Wheelchair Capacity scoring from 0 (dependent) to 3 (independent).
QUEST 2.0 - Usual Wheelchair | up to 4 weeks after enrollment
  The QUEST evaluates how satisfied one is with an assistive device.
QUEST 2.0 - Multispeed Wheelchair | up to 4 weeks after enrollment
  The QUEST evaluates how satisfied one is with an assistive device.

CONTACTS AND LOCATIONS:
Overall Officials: John M Looft, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Statistical Analysis Plan — https://osf.io/87wfq/files/osfstorage